CLINICAL TRIAL: NCT03989089
Title: Phase II, Single Arm, Open Label, Simon Two-Stage Study of Pembrolizumab in Metastatic HER2-negative Breast Cancer Patients: Evaluation of Impact of Germline Variants in APOBEC3B
Brief Title: Study of Pembrolizumab in Metastatic HER2-negative Breast Cancer Patients With APOBEC3B Mutation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Malaya (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National University Hospital, Singapore (Other); Cancer Research Malaysia (Other)
Responsible Party: Principal Investigator, Ho Gwo Fuang, Professor Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-UM2018001
Record Dates: First submitted 2019-02-25; First posted 2019-06-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: HER2-Negative Breast Cancer
Keywords: Germline APOBEC3B mutation; Pembrolizumab
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab single agent (Experimental): Pembrolizumab 200 mg will be given intravenously every 3 weeks , on Day 1 on each 3 week cycle. Pembrolizumab can be given up to 35 adminstration (2 years).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — The planned dose of pembrolizumab for this study is 200 mg every 3 weeks (Q3W). Based on the totality of data generated in the Keytruda® development program, 200 mg Q3W is the appropriate dose of pembrolizumab for adults across all indications and regardless of tumour type.
  All participants who off study treatment with stable disease (SD) or better may be eligible for up to an additional 17 cycles (approximately 1 year) of pembrolizumab treatment if they progress after stopping study treatment from the initial treatment phase. This retreatment is termed the Second Course Phase of this study and is only available if the study remains open and the participant met certain criteria as stated in the protocol.
  Other Names: Keytruda

SUMMARY:
This is an open label investigator initiated Phase II study of single agent pembrolizumab (Keytruda) in metastatic HER2-receptive negative breast cancer patients with germline deletion in the cytosine deaminase (APOBEC3B) gene. Approximately 44 subjects from Malaysia and Singapore will be enrolled in this study to examine the efficacy of pembrolizumab when given 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations (2 years). This study will be conducted in conformance with Good Clinical Practices. Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart.

DETAILED DESCRIPTION:
This is an open label investigator initiated Phase II study of single agent pembrolizumab (Keytruda®) in metastatic HER2-receptive negative breast cancer patients with germline deletion in the cytosine deaminase (APOBEC3B) gene. Approximately 44 subjects will be enrolled in this study to examine the efficacy of pembrolizumab when given 200 mg intravenously (IV) every 3 weeks (Q3W) for up to 35 administrations (2 years). ER+ patients need to have failed at least one line of prior hormonal treatment. All patients need to have failed at least one line, but no more than 3 lines, of prior chemotherapy in the metastatic setting.

Disease status will be followed by imaging studies at 9 weekly interval (± 7 days) during the first year, independent of any treatment delays, and every 12 weeks (±7 days) after the first year, until disease progression, start of non-study treatment, withdrawal of consent to study participation, death or end of the study. RECIST 1.1 will be used as the primary efficacy endpoint of response rate. Safety will be monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

Study treatment will continue until any of the following occurs:

1. Disease progression, as defined by Response Evaluation Criteria in Solid Tumour (RECIST version 1.1) (when progressive disease [PD] is confirmed, subject may be further followed up using consensus guideline of modified RECIST 1.1 [iRECIST] criteria);
2. Unacceptable toxicity;
3. Intercurrent illness that necessitates discontinuation of study treatment;
4. Investigator's decision to withdraw the subject,
5. Pregnancy;
6. Non-compliance with study treatment or procedure requirements;
7. Withdrawal of consent to treatment;
8. Death;
9. End of the study;
10. Other administrative reasons requiring cessation of study treatment.

This study will be conducted in conformance with Good Clinical Practices.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart - Section 6.0. Details of each procedure are provided in Section 7.0 - Trial Procedures.

Subject will be given a pre-screening inform consent form to participate in the genetic testing to determine their APOBEC3B germline mutation status.

Subject with confirmed APOBEC3B germline mutation will be given another inform consent form to participate in the main study.

The primary objective of the trial is to determine the efficacy of pembrolizumab in metastatic HER2-negative breast cancer subjects with APOBEC3B germline deletion polymorphism. Secondary objectives include progression-free survival (PFS), overall survival (OS) and response duration in this subject populations. The relationships of the germline variation, the associated molecular signatures, as well as other potential prognostic biomarkers with the study treatment will be explored as the exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed HER2-negative breast cancer (infiltrating ductal or lobular breast carcinoma) with measurable metastatic disease.
2. Must have received at least one but not more than three (3) prior lines of palliative chemotherapy for metastatic breast cancer.
3. Have received at least one line of hormonal therapy in the metastatic setting, for patients with ER+ (positive) breast cancer.
4. Documented germline APOBEC3B mutation (i.e. germline deletion).
5. Can provide archival tumour tissue sample or willing to provide tissues from a newly obtained core or excisional biopsy of a tumour lesion not previously irradiated. Note: Formalin-fixed, paraffin embedded (FFPE) tissue blocks or slides allowed (10 unstained slides are needed);
6. Have measurable disease based on RECIST 1.1 as determined by local radiology review. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (assessed within 10 days prior to the start of study treatment).
8. Have life expectancy of at least 3 months.
9. Have adequate organ function, within 10 days prior to the start of study treatment, as defined in the following:

   1. Absolute neutrophil count (ANC) ≥ 1,500/µl.
   2. Hemoglobin (Hb) ≥ 9 g/dL or 5.6mmol/La.
   3. Platelets > 100,000/µl.
   4. Creatinine ≤ 1.5 times ULN.
   5. ALT (SGPT) and AST (SGOT) ≤ 2.5 times the ULN (≤5 times for patients with liver metastases).
   6. Total bilirubin ≤ 1.5 mg/dL.
10. LDH ≤2.0 times the ULNWomen of child-bearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study treatment.
11. Women of child-bearing potential prepared to use adequate contraceptive measures if sexually active for the course of the study through 120 days after the last dose of treatment.
12. Have signed informed consent and able to comply with scheduled visits, treatment plan and other study procedures.

Exclusion Criteria:

1. Has HER2-positive breast cancer (FISH/CISH confirmed status, or 3+ IHC status)
2. Has use of any investigational agent or participation in another therapeutic clinical trial concurrently or in the 30 days prior to inclusion.
3. Has not recovered (e.g. to ≤Grade 1 or to baseline) from AEs due to a previously administrated therapy. Note: Participants with ≤Grade 2 neuropathy may be eligible.
4. Has an active autoimmune disease that has required systemic treatment in the past 2 years (e.g. with the use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systematic treatment.
5. Has a diagnosis of immunodeficiency or is receiving systematic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study treatment.
6. Has a concurrently active second malignancy, other than adequately treated non-melanoma skin cancers, in situ melanoma or in situ cervical cancer. Subjects with other non-mammary malignancies must have been disease-free for at least 5 years.
7. Has known active CNS metastases and/or carcinomatous meningitis. Previously treated brain metastases may participate provided these remain stable.
8. Has received prior therapy with an anti-PD1, anti-PDL1 or anti-PDL2 agent or with an agent directed to another co-inhibitory T cell receptor (such as CTLA-4, OX-40, and CD137) or has previously participated in pembrolizumab clinical studies.
9. Patient who has received a live vaccine within 30 days of the first dose of study drug.
10. Known hypersensitive or allergy to pembrolizumab and any of its components.
11. Patient who is pregnant or breastfeeding.
12. Patient with an expected life expectancy of less than 3 months.
13. History of significant comorbidities that, in the opinion of the investigator, may interfere with the conduct of the study, the evaluation of response, or with informed consent.
14. Active uncontrolled infection at the time of inclusion.
15. Has a history of class II-IV congestive heart failure or myocardial infraction.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of this study
17. Has evidence of active pneumonitis, or non-infectious pneumonitis requiring treatment with steroids.
18. Has a known history of Human Immunodeficiency Virus (HIV).
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on gender identity.
Enrollment: 44 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 4 years
  To determine the overall response rate (ORR) to the pembrolizumab treatment in metastatic HER2-negative breast cancer patients with germline APOBEC3B deletion polymorphisms using RECIST 1.1.

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 4 years
  To estimate the progression free survival (PFS) to the pembrolizumab treatment in metastatic HER2-negative breast cancer patients with germline APOBEC3B deletion polymorphisms.
Overall survival | Up to 4 years
  To estimate overall survival (OS) to the pembrolizumab treatment in metastatic HER2-negative breast cancer patients with germline APOBEC3B deletion polymorphisms.
Disease control rate | Up to 4 years
  To estimate the disease control rate (DCR) i.e. complete response (CR), partial response (PR) or stable disease (SD) to the pembrolizumab treatment in metastatic HER2-negative breast cancer patients with germline APOBEC3B deletion polymorphism.

CONTACTS AND LOCATIONS:
Overall Officials: Adlinda Alip, FRCR, Principal Investigator — University of Malaya
Locations (2):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Ho GF, Lee SC, Bustam AZ, Alip A, Abdul Satar NF, Saad M, Malik RA, Lim SE, Ow SGW, Wong A, Chong WQ, Ang YLE, Lee AWY, Hasan SN, Tuan Zaid N, Law KB, Toh YY, Tan HC, Selvam B, Lim J, Pan JW, Teo SH. Pembrolizumab monotherapy for previously treated metastatic HER2-negative breast cancer with germline APOBEC3B deletion: results of the phase II AUROR study. Lancet Reg Health West Pac. 2025 Jul 13;60:101637. doi: 10.1016/j.lanwpc.2025.101637. eCollection 2025 Jul. PMID 40697533